CLINICAL TRIAL: NCT07153510
Title: "Comparison of Post-Isometric Relaxation and Active Static Stretching Technique in Improving Hamstring Flexibility Among Allied Health Sciences Students"
Brief Title: "Comparative Effects of PIR and Static Stretching on Hamstring Flexibility" Post-Isometric Relaxation
Acronym: PIR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Tooba Arif, Dr. Tooba Arif, PT, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHS/DPS-25/1189
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hamstring Tightness; Hamstring Flexibility
Keywords: Hamstring tightness,; Post Isometric Relaxation; Active Static Stretching; Students; Allied Health Sciences
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-Isometric Relaxation (Experimental): Participants will undergo Post-Isometric Relaxation technique targeting the hamstring muscles. The technique involves an isometric contraction of the hamstring followed by a passive stretch. Participant will be in supine position; hip at 90° flexion, Isometric contraction of hamstrings for 7 seconds, Followed by 15 seconds of passive stretch, 10 repetitions, 3 times/week for 4 weeks
  Interventions: Other: Post-Isometric Relaxation
- Active Static Stretching (Experimental): Participants will perform Active Static Stretching exercises for the hamstrings, where the stretch is held actively without assistance.Seated long sitting position. Participant actively stretches hamstrings for 30 seconds. 10 repetitions, 3 times/week for 4 weeks
  Interventions: Other: Active Static Stretching

INTERVENTIONS:
Other: Post-Isometric Relaxation — Participants will undergo Post-Isometric Relaxation technique targeting the hamstring muscles. The technique involves an isometric contraction of the hamstring followed by a passive stretch. Participant will be in supine position; hip at 90° flexion, Isometric contraction of hamstrings for 7 seconds, Followed by 15 seconds of passive stretch, 10 repetitions, 3 times/week for 4 weeks
  Arms: Post-Isometric Relaxation
Other: Active Static Stretching — Participants will perform Active Static Stretching exercises for the hamstrings, where the stretch is held actively without assistance.Seated long sitting position. Participant actively stretches hamstrings for 30 seconds. 10 repetitions, 3 times/week for 4 week
  Arms: Active Static Stretching

SUMMARY:
Hamstring tightness is a common problem among students and young adults, often leading to reduced flexibility, musculoskeletal discomfort, and risk of injury. Different stretching methods are used in physiotherapy practice to improve muscle length and flexibility. Post-Isometric Relaxation (PIR), a type of muscle energy technique, and Active Static Stretching (ASS) are two commonly applied methods, but evidence comparing their effectiveness in improving hamstring flexibility among Allied Health Sciences students remains limited.

This randomized controlled trial aims to compare the effects of PIR and Active Static Stretching on hamstring flexibility in healthy university students. Participants will be randomly assigned to either PIR or ASS groups and undergo stretching sessions for a specified duration. Hamstring flexibility will be measured using the Active Knee Extension test before and after the intervention. The findings will provide evidence to guide physiotherapy education and clinical practice on the most effective stretching technique for improving hamstring flexibility.

DETAILED DESCRIPTION:
Hamstring muscle tightness is one of the most common musculoskeletal concerns in young adults, particularly in students of Allied Health Sciences who often spend prolonged hours in sitting postures during academic activities. Reduced hamstring flexibility is associated with altered posture, restricted range of motion, musculoskeletal discomfort, and a higher risk of lower limb injuries. Stretching interventions are widely used to address muscle tightness, with Post-Isometric Relaxation (PIR) and Active Static Stretching (ASS) being among the most frequently applied techniques in physiotherapy practice.

Post-Isometric Relaxation (PIR) is a form of muscle energy technique that utilizes a submaximal isometric contraction of the target muscle followed by a passive stretch, aiming to induce reflex relaxation and elongation of the muscle. Active Static Stretching (ASS) involves actively holding the muscle in a lengthened position for a fixed duration, relying on voluntary control and sustained tension to improve flexibility. While both techniques are clinically relevant, comparative evidence regarding their relative effectiveness in improving hamstring flexibility among young healthy populations, particularly Allied Health Sciences students, remains limited.

This randomized controlled trial is designed to compare the immediate and short-term effects of PIR and ASS on hamstring flexibility. A total of 54 students who meet the inclusion criteria will be randomly allocated to either the PIR group or the ASS group. Each group will undergo a structured stretching protocol for a specified period under supervision. Hamstring flexibility will be evaluated pre- and post-intervention using the Active Knee Extension (AKE) test, a valid and reliable measure of hamstring length.

The results of this study are expected to provide evidence on whether PIR or ASS is more effective for improving hamstring flexibility in this population. Findings will have important implications for physiotherapy education, clinical decision-making, and injury prevention strategies in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-25 years, Active Knee Extension (AKE) test angle > 20°, Willing to participate and provide informed consent

Exclusion Criteria:

* Any history of hamstring strain or lower limb injury in the past 6 months, Neurological or musculoskeletal disorders, Participation in other flexibility or stretching programs

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Hamstring flexibility | 4 weeks
  Hamstring flexibility, assessed by the Active Knee Extension (AKE) test using a universal goniometer.
  Assessment Timeline:
  Baseline (Day 0) Post-intervention (End of Week 4)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Lahore, Punjab Province, Pakistan